CLINICAL TRIAL: NCT02615899
Title: Effectiveness of Impairment Specific Exercises for Balance and Fall Risk in Community-Living Older Adults at Risk: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Sheri Silfies, Associate Professor, Research Lab Coordinator, Department of Physical Therapy & Rehabilitation Sciences, Drexel University, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1305002061
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Balance, Postural; Exercise Therapy
Keywords: Older Adults, Falls

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Matched (Active Comparator): Administer Targeted (specific) balance exercise interventions
  Interventions: Other: Matched: Targeted (specific) balance exercise interventions
- Mismatched (Active Comparator): Administer Untargeted (non-specific) balance exercise interventions
  Interventions: Other: Mismatched: Untargeted (non-specific) balance exercise interventions

INTERVENTIONS:
Other: Matched: Targeted (specific) balance exercise interventions
  Arms: Matched
Other: Mismatched: Untargeted (non-specific) balance exercise interventions
  Arms: Mismatched

SUMMARY:
Background Balance impairment is a key factor contributing to falls in older adults. Conceptually, clinicians may be able to prescribe targeted exercises if specific impairments can be identified. Objective Our objective was to use a model of balance subsystems to identify balance impairments and demonstrate the effectiveness of targeted (matched) exercises to improve balance and reduce fall risk in community-dwelling older adults. The investigators used the Balance Evaluation System Test (BESTest) as the model because it categorizes balance into 6 subsystems. Design Randomized, partially blinded, pretest-post-test clinical trial consisting of 2 Phases: 1. A comparison between impairment-matched exercises and a control, and 2. A comparison between impairment-matched and mismatched exercises. Setting Senior independent living community. Participants Adult volunteers (n = 40; aged 74-94) recruited as sample of convenience who met the criteria. Participants (n = 20) identified with impairment in the biomechanical (BC) constraints subsystem and participants (n = 20) with impairment in anticipatory postural adjustment (APA) subsystem were enrolled and randomized into 2 subgroups (matched and control/delayed mismatched; n = 10 each subgroup). Intervention Phase 1: Participants in the matched subgroup received a 6-week exercise program matched to their impaired subsystem while the mismatched subgroup served as control. Phase 2: Following the delay, participants in the mismatched group received a 6-week exercise program mismatched to their impairment. Measurements Primary outcome variables were scores on the targeted subsystem (BC, APA), BESTest total, Berg Balance Scale, and fear of falling measure. Quality of life was a secondary outcome. Outcome data were collected by the tester blind to pretest scores and group allocation. Results The matched exercise subgroups demonstrated both statistical and clinical improvement in all outcome variables compared to the control; and showed greater improvement in balance impairments compared to the mismatched subgroup, but not in fall risk reduction. Limitations The therapist who administered the pretest knew the subgroup assignment and implemented the exercises. Conclusions Results provide preliminary evidence that using a balance assessment model to identify impairments in the BC and APA subsystems and prescribing targeted exercises reduces these balance impairments for older adults and may warrant future studies.

ELIGIBILITY:
Inclusion Criteria:

* individuals who met the criteria for a concurrent psychometric study (older adults aged 65 years and older, cognitively able to understand and follow simple instructions,and able to walk independently with or without an assistive device for more than 100 ft); and demonstrated
* elevated fracture risk
* elevated fall risk
* impaired balance in either the BC or APA subsystem of balance as identified with BESTest.

Exclusion Criteria:

* individuals who had:

  * a progressive diseases or unstable medical conditions
  * major surgery in the past 3 months
  * physician's orders not to participate in an exercise program for any reason
  * impairment in both BC and APA subsystems
  * impairments in more than a total of 3 subsystems
  * who were currently receiving treatment for balance or fall prevention.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
BESTest total | 6 weeks
  Balance
Targeted subsystem of BESTest (APA or BC subsystem) | 6 weeks
  Subsystem balance
Berg Balance Scale | 6 weeks
  Fall risk indicator
the University of Illinois at Chicago Fear of Falling Measurement (UIC FFM) | 6 weeks
  Fall risk indicator

SECONDARY OUTCOMES:
Short Form Health Survey (SF-12, Version 2; QualityMetric Inc.) questionnaire | 6 weeks
  Quality of Life indicator

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Smith, PT, PhD, Study Chair — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States